CLINICAL TRIAL: NCT06301308
Title: A Novel Application of 2% Lidocaine Injection for Male Rigid cycstoscopy-a Patient-blinded Randomised Trial
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The standard measures of anaesthesia in cystoscopy are not uniform internationally, and given this, we were unable to recruit the first participant in the study.
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Cheng Shunhua, Co-chief superintendent nurse, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022021
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Lidocaine; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intraurethral lidocaine gel alone (Sham Comparator): Participants received 10 ml of intraurethral lidocaine gel at a concentration of 2%
  Interventions: Drug: Intraurethral lidocaine gel alone
- Intraurethral lidocaine gel + lidocaine 2% injection (Experimental): Participants received 10 ml of intraurethral lidocaine gel at a concentration of 2% and using the injection of lidocaine 2% to irrigate the urethra using a 20 ml syringe.
  Interventions: Drug: Intraurethral lidocaine gel + lidocaine 2% injection
- intraurethral lidocaine gel + liquid paraffinl (Experimental): Liquid paraffin were used to lubricate hte cystoscopy tube AND participants received 10 ml of intraurethral lidocaine gel at a concentration of 2%
  Interventions: Drug: intraurethral lidocaine gel + liquid paraffinl

INTERVENTIONS:
Drug: Intraurethral lidocaine gel alone — participants received 10 ml of intraurethral lidocaine gel at a concentration of 2%
  Other Names: Group A
  Arms: Intraurethral lidocaine gel alone
Drug: Intraurethral lidocaine gel + lidocaine 2% injection — participants received 10 ml of intraurethral lidocaine gel at a concentration of 2% and using the injection of lidocaine 2% to irrigate the urethra using a 20 ml syringe.
  Other Names: Group B
  Arms: Intraurethral lidocaine gel + lidocaine 2% injection
Drug: intraurethral lidocaine gel + liquid paraffinl — Liquid paraffin were used to lubricate hte cystoscopy tube AND participants received 10 ml of intraurethral lidocaine gel at a concentration of 2%
  Other Names: Group C
  Arms: intraurethral lidocaine gel + liquid paraffinl

SUMMARY:
The goal of this clinical trial is to learn about a novel application of lidocaine injection in male patients who needs rigid cycstoscopy test. The main question it aims to answer is:Does New Application of Lidocaine Liquid Provide Pain Relief for Patients During Cystoscopy? Before the cycstoscopy,Participants will be randomly divided into three different anesthesia mode groups,namely are Group A (intraurethral lidocaine gel alone), Group B (intraurethral lidocaine gel + lidocaine 2% injection), and Group C (intraurethral lidocaine gel + liquid paraffinl).Patients only need to prepare and cooperate according to routine surgical operations，which is group B or group C.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to investigate the efficacy of a novel application of lidocaine injection in alleviating pain for male patients undergoing rigid cystoscopy procedures. Rigid cystoscopy is a common diagnostic examination used to visualize the interior of the bladder and urethra. However, it can be associated with discomfort and pain for patients.

The central question driving this study is whether the new application of lidocaine liquid can provide effective pain relief during cystoscopy. To address this question, participants will be randomly assigned to one of three anesthesia mode groups: Group A, which will receive intraurethral lidocaine gel alone; Group B, which will receive intraurethral lidocaine gel along with lidocaine 2% injection; and Group C, which will receive intraurethral lidocaine gel along with liquid paraffin.

Those assigned to Group B or Group C will only need to prepare and cooperate according to routine surgical operations. This standardizes the pre-procedural preparation process across the study groups, ensuring consistency in the approach to anesthesia administration.

By comparing the pain levels experienced by patients in each group during cystoscopy, the study aims to determine the effectiveness of the new lidocaine application method in providing pain relief. This information will be crucial in improving the patient experience during cystoscopy procedures and potentially optimizing anesthesia protocols for future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male patients under the age of 50 referred for postoperative cystoscopy for bladder cancer

Exclusion Criteria:

- 1. Other evident causes contributing to lower urinary tract symptoms, such as obvious glandular cystitis and severe urinary tract infections.

2. Excessive prostatic hyperplasia. 3. Urethral stricture. 4. A history of prior urethral surgeries. 5. Uncontrolled hypertension, cardiac conditions, and chronic obstructive pulmonary disease.

Max Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Access the pain score using the Visual Analogue Scale (VAS) | The procedure was evaluated using the visual analogue scale immediately afterward (referred to as "during the procedure" for the study's purposes) and again five minutes later.
  Access the pain score assessed using the Visual Analogue Scale (VAS) during the procedure

SECONDARY OUTCOMES:
Postoperative complications | Within three days after surgery.
  The second outcomes were included parameters such as field of view occlusion, duration of pain, hematuria duration, and lower urinary tract symptoms post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shunhua Cheng, Study Chair — Central South University,the second xiangya hospital; Can Tang, Study Director — Central South University,the second xiangya hospital; Shunhua Cheng, Principal Investigator — Central South University,the second xiangya hospital
Locations (1):
- The second xiangya hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT06301308/Prot_SAP_ICF_000.pdf